CLINICAL TRIAL: NCT00228293
Title: Assessment of Cardiopulmonary Resuscitation Quality During In-Hospital Cardiac Arrest
Brief Title: Assessing CPR Quality During In-Hospital Cardiac Arrest
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB11754B; IDE G020121
Record Dates: First submitted 2005-09-23; First posted 2005-09-28 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; CPR
MeSH Terms: conditions — Heart Arrest | interventions — Defibrillators

INTERVENTIONS:
Device: investigational monitor/defibrillator with CPR feedback

SUMMARY:
Using an investigational monitor/defibrillator that passively records CPR quality parameters, including chest compression rate and depth and ventilation rate and volume, we are prospectively recording CPR quality during sequential in-hospital cardiac arrests at the University of Chicago Hospitals. Using an audio feedback system linked to this device, we are studying whether such audio feedback improves CPR quality when provided to rescuers trained in the use of the device.

DETAILED DESCRIPTION:
Patients who suffer cardiac arrest during their hospitalization at the University of Chicago hospitals are given CPR and other resuscitation measures by trained physician and nurse teams. This care is given with the use of defibrillators to monitor cardiac rhythm as well as provide defibrillation as needed.

We have worked closely with engineers at Laerdal Medical Corporation to develop a defibrillator that passively monitors the quality of CPR via additional external sensors (see details in the following reference: Abella BS, Alvarado JP, Myklebust H, Edelson DP, Barry A, O'Hearn N, Vanden Hoek TL, Becker LB. Quality of cardiopulmonary resuscitation during in-hospital cardiac arrest. JAMA. 2005;293:305-10).

Patients who suffer in-hospital arrest are enrolled (provided they are over 16 years of age, are not pregnant, and are not in the operating room or emergency room setting) with mechanisms to satisfy IRB waiver of consent provisions. These patients receive the same care as before the study, but CPR parameters are recorded by the device. In addition, the device provides audio/visual "coaching" in CPR, based on the actual performance of CPR as measured.

We hypothesize that this coaching will improve CPR quality and hopefully improve survival from cardiac arrest.

The first phase of investigation is now complete, where patients were enrolled and studied without feedback ("baseline" group). Now we are enrolling patients into a second group with feedback provided. Enrollment is nearly complete for this second group. We will then evaluate the baseline and feedback groups to ascertain whether CPR improved over the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with cardiac arrest hospitalized at University of Chicago Hospitals

Exclusion Criteria:

* pregnant
* arrest in ER or OR
* pediatric patient
* patient DNR, no CPR given
* no CPR given for other reasons (e.g. shock only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-12; Study Completion 2005-09

PRIMARY OUTCOMES:
parameters of CPR quality:
chest compression rate
chest compression depth
ventilation rate
ventilation depth
CPR pause times

SECONDARY OUTCOMES:
return of spontaneous circulation (ROSC)
survival to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lance B Becker, MD, Principal Investigator — Professor of Medicine, University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States

REFERENCES:
- [Result] Abella BS, Alvarado JP, Myklebust H, Edelson DP, Barry A, O'Hearn N, Vanden Hoek TL, Becker LB. Quality of cardiopulmonary resuscitation during in-hospital cardiac arrest. JAMA. 2005 Jan 19;293(3):305-10. doi: 10.1001/jama.293.3.305. PMID 15657323
- [Derived] Edelson DP, Litzinger B, Arora V, Walsh D, Kim S, Lauderdale DS, Vanden Hoek TL, Becker LB, Abella BS. Improving in-hospital cardiac arrest process and outcomes with performance debriefing. Arch Intern Med. 2008 May 26;168(10):1063-9. doi: 10.1001/archinte.168.10.1063. PMID 18504334
- [Derived] Kramer-Johansen J, Edelson DP, Abella BS, Becker LB, Wik L, Steen PA. Pauses in chest compression and inappropriate shocks: a comparison of manual and semi-automatic defibrillation attempts. Resuscitation. 2007 May;73(2):212-20. doi: 10.1016/j.resuscitation.2006.09.006. Epub 2007 Jan 22. PMID 17241734